CLINICAL TRIAL: NCT00798694
Title: Ocular Surface Changes With Topical Prostaglandin Analog Therapy
Brief Title: How Similar Are Changes to the Surface of the Eye When Two Different Glaucoma Eye Drops Are Used?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, L. Jay Katz MD, Principal Investigator, Wills Eye
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-875
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Glaucoma
Keywords: glaucoma; impression cytology; ocular surface changes; prostaglandins
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost; Prostaglandins, Synthetic; Travoprost

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Doctors assessing patients were masked to treatment. Patients used open label Xalantan in the right eye and Travatan Z in the left eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- New to Meds (Other): Naive to glaucoma therapy medical or surgical. All patients will receive Xalatan in the right eye and Travatan Z in the left eye.
  Interventions: Drug: Xalatan; Drug: Travatan Z
- Currently on Xalatan (Other): Patients currently on Xalatan at least one month. All patients will receive Xalatan in the right eye and Travatan Z in the left eye.
  Interventions: Drug: Xalatan; Drug: Travatan Z

INTERVENTIONS:
Drug: Xalatan — one drop of Xalatan Ophthalmic Solution instilled in right eye at bedtime
  Other Names: prostaglandin analog
Drug: Travatan Z — one drop of Travatan Z Ophthalmic Solution instilled in left eye at bedtime
  Other Names: prostaglandin analog

SUMMARY:
To determine whether one glaucoma eye drop is less likely to cause changes to the surface of the eye (conjunctiva) than another. The two different prostaglandins are Xalatan and Travatan Z.

DETAILED DESCRIPTION:
Two groups will be entered into this study: group 1 will be naive to treatment and group 2 will be using Xalatan for at least one month before enrollment. Both groups will be using one drop at bedtime of Xalatan in the right eye and one drop at bedtime of Travatan Z in the left eye. Both of these drops are presently on the market and approved by the FDA for treatment of lowering eye pressure. Because this study will be masked, the examining clinician will not know what study drop each patient has been using.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Able to understand protocol and agree to 3 visits
* Any type of glaucoma
* Selective laser trabeculoplasty, Argon laser trabeculoplasty, peripheral iridotomy accepted
* Naïve: No prior glaucoma treatment (medical or surgical)
* If patient non-compliant, must be off meds 3 months
* Xalatan: At least one month use

Exclusion Criteria:

* Both Groups: Any history of ocular surface disease
* Dry eye syndrome or prior Restasis use
* Prior ocular surgery other than cataract extractions
* Uveitis or other inflammatory disease of the eye or adnexa
* Systemic medications that might influence ocular inflammation
* Any active inflammation or infection
* Pregnancy or intention to become pregnant
* Naïve: Prior use of topical glaucoma medication unless off for 3 months.
* Use of preserved artificial tear preparations in last 30 days and more than one year history of chronic use
* Xalatan: Prior use of Travatan or Travatan Z

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie J Katz, MD, Principal Investigator — Wills Eye Glaucoma Service
Locations (1):
- Wills Eye Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
A manuscript has been published.

REFERENCES:
- [Result] Gupta SR, Ichhpujani P, Wizov SS, Wittpenn JR, Moster MR, Pro MJ, Rapuano CJ, Cruz-Colon C, Myers JS, Katz LJ. Effects of Latanoprost Versus Travoprost with Sofzia on Ocular Surface. ARVO E-abstract 168/A391 2010
- [Result] Rahmatnejad K, Rapuano CJ, Ichhpujani P, Wizov SS, Moster MR, Hark LA, Katz LJ. The Effects of Latanoprost With Benzalkonium Chloride Versus Travoprost With SofZia on the Ocular Surface. Eye Contact Lens. 2018 Nov;44 Suppl 2:S93-S98. doi: 10.1097/ICL.0000000000000405. PMID 28617732

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (New to Meds): Naive to glaucoma therapy medical or surgical. These patients have never used eye drops to lower eye pressure. All patients will receive Xalatan in the right eye and Travatan Z in the left eye.
  Xalatan: one drop of Xalatan Ophthalmic Solution instilled in right eye at bedtime
  Travatan Z: one drop of Travatan Z Ophthalmic Solution instilled in left eye at bedtime
- Group 2 (Currently on Xalatan): Patients currently on Xalatan at least one month. These patients have been using Xalatan at least one month to lower their eye pressure. All patients will receive Xalatan in the right eye and Travatan Z in the left eye.
  Xalatan: one drop of Xalatan Ophthalmic Solution instilled in right eye at bedtime
  Travatan Z: one drop of Travatan Z Ophthalmic Solution instilled in left eye at bedtime
Period: Overall Study
Arm/Group | Group 1 (New to Meds) | Group 2 (Currently on Xalatan)
Started | 30 | 28
Completed | 28 | 27
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: 58 patients were enrolled. 2 patients did not return for follow-up and 1 patient's intraocular pressure was not controlled adequately on one eye drop. That patient was discontinued when a second eye drop was added to lower their eye pressure.
Groups:
- Group 1 (New to Meds): Naive to glaucoma therapy medical or surgical. All patients will receive Xalatan in the right eye and Travatan Z in the left eye.
  Xalatan: one drop of Xalatan Ophthalmic Solution instilled in right eye at bedtime
  Travatan Z: one drop of Travatan Z Ophthalmic Solution instilled in left eye at bedtime
- Group 2 (Currently on Xalatan): Patients currently on Xalatan at least one month. All patients will receive Xalatan in the right eye and Travatan Z in the left eye.
  Xalatan: one drop of Xalatan Ophthalmic Solution instilled in right eye at bedtime
  Travatan Z: one drop of Travatan Z Ophthalmic Solution instilled in left eye at bedtime
- Total: Total of all reporting groups
Arm/Group | Group 1 (New to Meds) | Group 2 (Currently on Xalatan) | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.7) | 61.2 (13.2) | 61.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 15 | 11 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 15 | 17 | 32
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Change in Tear Break up Time (TBUT)
Description: Difference of tear break up time (in seconds, average of 3 measurements) at one and two months after enrollment.
Time Frame: Baseline, 1 month, 2 months
Population: Both eyes combined change from baseline.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- New to Meds: Naive to glaucoma therapy medical or surgical. All patients will receive Xalatan in the right eye and Travatan Z in the left eye.
  Xalatan: one drop of Xalatan Ophthalmic Solution instilled in right eye at bedtime
  Travatan Z: one drop of Travatan Z Ophthalmic Solution instilled in left eye at bedtime
  A geometric mean ratio of 1 indicates equivalence of the two geometric means.
Arm/Group | New to Meds | Currently on Xalatan
Number analyzed (Participants) | 28 | 27
seconds
  1 month | -0.86 (6.09) | -0.59 (4.70)
  2 months | -2.00 (5.42) | 0.27 (4.72)
Statistical Analysis 1: Comparison: New to Meds vs Currently on Xalatan; Null Hypothesis: There is no significant difference in tear break-up time between the group "New to Meds" and the group "Currently on Xalatan" at two months; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Tear Production
Description: Tear production, measured by Schirmer test in millimeters
Time Frame: Baseline, 1 month, 2 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Group 1 (New to Meds) | Group 2 (Currently on Xalatan)
Number analyzed (Participants) | 28 | 27
millimeters
  Baseline | 22.4 (8.7) | 17.1 (9.3)
  1 month | 21.1 (9.6) | 17.4 (9.0)
  2 months | 23.0 (9.35) | 17.4 (9.8)

3. Secondary Outcome: Conjunctival Hyperemia Score
Description: Conjunctival hyperemia is the amount of redness on the white part of the eye. A total score was obtained by the sum of assessments in 6 areas of each eye are which are scored from 0 to 3 (0 = no redness; 3 = severe redness), then summed per eye for a total score range of 0-18 (0 = no redness; 18 = severe redness).
Time Frame: Baseline, 1 month, 2 months
Population: One eye per participant in each Arm
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1 Xalatan: 28 patients - Eye using Xalatan (latanoprost with benzalkonium chloride)
- Group 1 Travatan Z: 28 patients - Eye using Travatan Z (travoprost with SofZia)
- Group 2 Xalatan: 27 patients - Eye using Xalatan (latanoprost with benzalkonium chloride)
- Group 2 Travatan Z: 27 patients - Eye using Travatan Z (travoprost with SofZia)
Arm/Group | Group 1 Xalatan | Group 1 Travatan Z | Group 2 Xalatan | Group 2 Travatan Z
Number analyzed (Participants) | 28 | 28 | 27 | 27
units on a scale
  Baseline | 4.0 (2.7) | 4.6 (3.3) | 3.2 (2.6) | 3.6 (3.2)
  1 month | 4.0 (2.7) | 4.6 (3.3) | 3.4 (2.5) | 4.8 (3.2)
  2 months | 4.0 (3.5) | 5.3 (3.7) | 3.3 (3.3) | 4.0 (3.8)

4. Secondary Outcome: Intraocular Pressure
Description: Intraocular pressure (the fluid pressure inside the eye) was measured two times in each eye using the Goldman applanation tonometer and averaged.
Time Frame: Baseline, 1 month, 2 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group 1 Xalatan | Group 1 Travatan Z | Group 2 Xalatan | Group 2 Travatan Z
Number analyzed (Participants) | 28 | 28 | 27 | 27
mmHg
  Baseline | 20.9 (7.1) | 20.1 (6.3) | 14.8 (2.7) | 15.0 (3.3)
  1 month | 15.6 (3.8) | 15.5 (3.4) | 15.1 (2.8) | 14.5 (2.8)
  2 months | 14.6 (3.7) | 15.2 (3.8) | 14.6 (3.3) | 14.3 (3.3)

5. Secondary Outcome: Ocular Surface Disease Index Score
Description: Ocular Surface Disease Index Scores (OSDI) were obtained from a 12-item validated OSDI questionnaire completed by each participant. This is an assessment related to eye comfort. Each question's score ranges from 0 = no disability to 4 = greatest disability. The total score is multiplied by 25 then divided by the number of questions answered then matched to a grid ranging from 0 to 100 with 0 having symptoms reported none of the time versus 100 having disability symptoms reported all of the time.
Time Frame: Baseline, 1 month, 2 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group 1 Xalatan | Group 1 Travatan Z | Group 2 Xalatan | Group 2 Travatan Z
Number analyzed (Participants) | 28 | 28 | 27 | 27
scores on a scale
  Baseline | 10.8 (14.7) | 11.7 (14.2) | 9.8 (11.4) | 14.2 (17.7)
  1 month | 10.8 (14.7) | 11.7 (14.2) | 7.0 (6.9) | 8.1 (7.7)
  2 months | 11.1 (11.9) | 11.8 (11.6) | 6.6 (8.7) | 11.2 (18.3)

6. Secondary Outcome: Corneal Staining Score
Description: Corneal staining is an indication of the amount of dryness of the cornea (front clear part of the eye). A total score was obtained by the sum of assessments in five areas of each eye which are scored from 0 to 3 (0 = no dryness; 3 = severe dryness), then summed per eye for a total score range of 0-15 (0 = no dryness; 15 = severe dryness).
Time Frame: Baseline, 1 month, 2 months
Population: One eye from each patient per arm.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Group 1 Xalatan | Group 1 Travatan Z | Group 2 Xalatan | Group 2 Travatan Z
Number analyzed (Participants) | 28 | 28 | 27 | 27
scores on a scale
  Baseline | 0.7 (1.0) | 0.8 (1.0) | 1.0 (1.9) | 1.0 (1.8)
  1 month | 0.7 (1.0) | 0.8 (1.0) | 1.3 (2.0) | 1.2 (1.6)
  2 months | 1.0 (2.0) | 1.3 (1.9) | 1.0 (1.5) | 1.0 (0.9)

ADVERSE EVENTS:
Time Frame: Baseline, 1 month, 2 months
Arm/Group | New to Meds | Currently on Xalatan
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 0/30 | 0/28

LIMITATIONS AND CAVEATS:
Small sample size. Short term study may not reflect long term ocular surface. Patients selected were free of baseline Ocular Surface Disease (OSD). Sample population with pre-existing OSD may have different sensitivity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No